CLINICAL TRIAL: NCT01184144
Title: Effect of Pioglitazone on Peritoneal Cytokines in Women With Endometriosis
Brief Title: Endometriosis: Immunomodulation
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2010-0066
Record Dates: First submitted 2010-08-13; First posted 2010-08-18 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2012-04

CONDITIONS: Endometriosis
Keywords: Endometriosis; Peritoneal fluid; Cytokines; Peroxisome Proliferator-Activated Receptors
MeSH Terms: conditions — Endometriosis | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pioglitazone (Experimental): Pioglitazone study drug
  Interventions: Drug: Pioglitazone
- No drug (No Intervention): "Placebo" like comparitor

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone, 30 mg, by mouth daily for 2 weeks
  Other Names: Actos
  Arms: pioglitazone

SUMMARY:
The purpose of this study is to compare the effect of pioglitazone versus no drug on soluble profinflammatory markers in peritoneal fluid of women with endometriosis.

DETAILED DESCRIPTION:
The overall goal of this proposal is to assess modulation of immune mechanisms in endometriosis. Endometriosis is a common ailment affecting approximately five million reproductive-aged American women. We will test the efficacy of a novel immunomodulatory drug (peroxisome proliferator activated receptor gamma, PPAR-gamma, agonist), pioglitazone, to reduce peritoneal fluid cytokine concentrations in women with endometriosis compared with the non-treated controls (randomized controlled trial). Based on prior studies done by the investigator highlighting the major role of cytokines and the immune system in the genesis or propagation of endometriosis, these experiments could lead to improved translational treatment strategies and a better understanding of endometriosis. Acting through PPAR-gamma, TZDs inhibit proinflammatory cytokines as well as NF-kB, an important nuclear transcription factor for the production of many cytokines. Accordingly, since human endometrial epithelial and stromal cells contain PPAR-gamma, we felt i would be useful to evaluate the influence of a PPAR-gamma ligand, pioglitazone, on the concentration of specific peritoneal fluid cytokines.

Comparison: After the pre-trial screening, eligible subjects with presumed endometriosis and age 18-45 will be consented and randomly assigned to receive either pioglitazone (30 mg, daily)or no drug for 2 weeks. Peritoneal fluid will be collected at the time of surgery and the volume measured. All patients enrolled in the study will have their surgery during the follicular phase of the cycle in order to minimize differences in volume and cytokine concentration due to the cyclical changes. The primary measure will be the peritoneal fluid concentration comparisons of the two groups assessing six different cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy woman age 18 - 45 years.
2. Regular cycles (24-35 days).
3. Pelvic pain ≥ 3 months.
4. Negative pregnancy test.
5. Non-lactating.
6. No prior (<3 months) use of hormonal therapy.
7. No history of liver disease.
8. Suspected endometriosis and scheduled for surgery to confirm this diagnosis
9. Surgery scheduled in follicular phase.
10. Consent to participate in the study.
11. Enrollment into data analysis portion of study if:

    * Endometriosis diagnosed from surgical specimen by routine hematoxylin and eosin staining and histological evaluation.

Exclusion Criteria:

1. Major psychiatric conditions or the abuse of alcohol or drugs which would make it difficult for the subject to complete study procedures.
2. Active or prior infection with hepatitis, human immunodeficiency virus (HIV) infection, or history of high-risk activities (e.g., IV drug abuse) which would increase risk to laboratory personnel. Of note, no testing for hepatitis or HIV will be performed as part of this study and all tissues will be handled and discarded as if they were potentially infected.
3. Patients with liver dysfunction (elevated liver enzymes > 2 times the upper limit of normal).
4. Presence of pre-existing malignancy, including carcinoma of the breast or uterus.
5. Women with other causes of chronic pelvic pain including infectious, gastrointestinal, musculoskeletal, neurologic or psychiatric.
6. Elevated WBC.
7. NYHA functional class I-IV heart failure.
8. Diabetes mellitus.
9. Known pregnancy or positive pregnancy test.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Peritoneal cytokine levels | Within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dan I Lebovic, MD, Principal Investigator — Univ Wisconsin